CLINICAL TRIAL: NCT04150692
Title: ESCALADARA: Escalation of Daratumumab Frequency Following Biochemical Progression in Relapsed/Refractory Multiple Myeloma
Brief Title: Escalation of Daratumumab Frequency Following Biochemical Progression in Relapsed/Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Washington University School of Medicine (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201910200
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Dara-SC Re-Escalation (Experimental): -Re-escalation will include weekly dosing for two 4-week cycles (8 doses, Days 1, 8, 15, and 22 of each 28-day cycle) followed by dosing every-other-week thereafter (Days 1 and 15 of each 28-day cycle). Patients will remain on study treatment until meeting clinical progression.
  Interventions: Biological: Dara-SC; Procedure: Blood for research assessments; Procedure: Bone marrow for research assessments
- Arm 2: Dara-SC (Active Comparator): -Continued subcutaneous daratumumab and and hyaluronidase-fihj (1,800mg/30,000U, [Dara-SC])
  Interventions: Biological: Dara-SC; Procedure: Blood for research assessments; Procedure: Bone marrow for research assessments

INTERVENTIONS:
Biological: Dara-SC — -Subcutaneous daratumumab and hyaluronidase-fihj
Procedure: Blood for research assessments — -Cycle 1 Day 1, Cycle 3 Day 1, and at progression or end of study (whichever is first)
Procedure: Bone marrow for research assessments — -Cycle 1 Day 1, Cycle 3 Day 1, and at progression or end of study (whichever is first)

SUMMARY:
In a small case series, the investigators identified five patients who had an initial response to standard daratumumab (weekly for 2 cycles, every other week for 4 cycles, then monthly thereafter) either as mono- or combination therapy, who then had daratumumab frequency escalated when early biochemical progression was noted, an investigational endeavor. In this series, patients received a median of 5 additional cycles of daratumumab at an escalated frequency (range: 2-8). Additionally, the median change in involved paraprotein after one cycle of weekly-escalated dara was -40% (range: -67% to +5%), with most achieving prior partial response or stable disease.

In patients who initially have at least a partial response (PR) to daratumumab, who then have biochemical progression following de-escalation, it is conceivable that CD38 saturation is not optimized at the every 4 weeks dosing interval. The investigators believe that escalating the frequency of daratumumab in patients with biochemical progression, in this investigational setting, may recapture the initial response, delay clinical progression, and/or delay treatment changes.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma diagnosis according to IMWG criteria
* Prior achievement of PR or better on standard daratumumab (single-agent or combination therapy)
* On daratumumab for at least 7 months, currently on once-monthly dosing
* Evidence of biochemical progression only, confirmed via two consecutive assessments.

The interval between labs would generally be 1 to 4 weeks, and the second set of labs may be the screening assessment. Biochemical progression is defined as an increase of > 25% from lowest response value in any one or more of the following:

* Serum M-component (the absolute increase must be > 0.5 g/dL)
* Urine M-component (the absolute increase must be > 200 mg/24 h)
* The difference between involved and uninvolved FLC levels (the absolute increase must be > 10 mg/dL; only in patients without measurable serum and urine M-protein levels)

  * Age ≥ 18 years
  * Eastern Cooperative Oncology Group (ECOG) performance status 0-2
  * Adequate bone marrow reserve, with ANC >1500 and Platelets >75k without transfusion or growth factors within 7 days prior to assessment
  * Adequate hepatic function, with AST and ALT ≤ 3.5 times the upper limit of normal and bilirubin ≤ 2 mg/dL
  * Creatinine clearance (CrCl) ≥ 15 mL/minute within 7 days prior to enrollment, either measured or calculated using a standard formula
  * HBV DNA Tests: Subjects who are positive for Anti-HBc or Anti-HBs will undergo testing for hepatitis B DNA by PCR. Subjects with serologic findings suggestive of HBV vaccination (Anti-HBs positivity as the only serologic marker) and a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR. During and following study treatment, subjects who have history of HBV infection will be closely monitored for clinical and laboratory signs of reactivation of HBV as specified in the Time and Events Schedule. Where required by local law, the results of HBV testing may be reported to the local health authorities.
  * Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Evidence of clinical progression/relapse over the 3 months prior to confirmed eligibility, based on centralized laboratory data performed at Washington University School of Medicine or radiographic data independently reviewed at Washington University School of Medicineas defined as:

  * Development of new soft tissue plasmacytomas or bone lesions
  * Definite increase in the size of existing plasmacytomas or bone lesions. A definite increase is defined as a 50% (and at least 1 cm) increase as measured serially by the sum of the products of the cross-diameters of the measurable lesion
  * Hypercalcemia (> 11.5 mg/dL) [2.65 mmol/L]
  * Decrease in hemoglobin of > 2 g/dL [1.25 mmol/L] not attributable to another cause as determined by investigator
  * Rise in serum creatinine by 2 mg/dL or more [177 mmol/L or more] not attributable to another cause as determined by investigator
* Evidence of myeloma with in the CNS
* Diagnosis of plasma cell leukemia
* Prior allergic reaction to daratumumab or medications used in the treatment backbone
* Interruption in daratumumab therapy for any reason in the preceding 6 months longer than 8 weeks.
* Pregnant or lactating females - woman and men of childbearing potential are required to employ an effective contraceptive method as outlined in the ICF
* Concurrent malignancy other than MM requiring active treatment excluding skin cancer managed with local therapy
* Compromised cardiovascular function defined as any of the following:

  * EKG evidence of acute ischemia;
  * EKG evidence of medically significant conduction system abnormalities;
  * history of myocardial infarction within the last 6 months;
  * unstable angina pectoris or cardiac arrhythmia; (history of Class 3 or Class 4 New York Heart Association congestive heart failure.
* Severe persistent asthma (FEV1<60% and/or daily symptoms) or severe COPD defined clinically or by historical pulmonary function tests with an FEV1 <50% predicted
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy)
* Any other clinically significant medical disease or condition that, in the judgement of the investigator, would prevent the participant from safely participating in the trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years following initiation of treatment (estimated to 3 years and 8 months)
  -Defined as the length of time between Cycle 1 Day 1 and progressive disease or death. Patients who are alive and progression-free or were lost to follow-up at the time of data analyses will be censored on the last known alive date.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 6 months following initiation of treatment
  -Defined as the proportion of patients with a partial response (PR) or better following first treatment with daratumumab following randomization, as defined by IMWG criteria
Proportion of patients on treatment following 3 cycles | Completion of cycle 3 by all enrolled patients (estimated to be 12 weeks)
Paraprotein change between Cycle 1 and Cycle 2 of treatment | From cycle 1 through cycle 2 (estimated to be 8 weeks)
Overall survival | Up to 2 years following treatment removal (estimated to be 2 years and 8 months)
  -Overall survival (OS) will be defined as time from Cycle 1 Day 1 to death due to any causes. Patients who are alive or were lost to follow-up at the time of data analyses will be censored on the last known alive date.
Duration of response (DOR) | Up to 3 years following initiation of treatment (estimated to be 3 years and 8 months)
  -Defined as the length of time between initial response with daratumumab following randomization and progressive disease (in responders).

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Schroeder, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu